CLINICAL TRIAL: NCT00553371
Title: Assessment of the Utility of CT Follow Up in the Long Term Follow Up of Patients With Metastatic Non Seminomatous Germ Cell Tumour (NSGCT)
Brief Title: Follow-up Evaluation Using CT Scans in Patients Who Have Been Treated For Metastatic Testicular Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000573199; ICR-RMH-NSGCT; EU-20770
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2007-10

CONDITIONS: Testicular Germ Cell Tumor
Keywords: stage II malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor
MeSH Terms: conditions — Testicular Germ Cell Tumor; Testicular Neoplasms

INTERVENTIONS:
Other: biomarker analysis
Procedure: computed tomography

SUMMARY:
RATIONALE: Learning about long-term effects in patients with testicular cancer may help doctors plan better treatment and follow-up care.

PURPOSE: This clinical trial is using CT scans to follow patients who have been treated for metastatic testicular cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the frequency of relapse or recurrent abnormalities detected by CT scan in patients on long-term follow-up for metastatic nonseminomatous germ cell tumour (NSGCT).
* To assess the utility of CT scan-assessment in these patients.
* To assess the prognostic factors predictive of late relapse in NSGCT.

OUTLINE: This is a multicenter study.

Patients are screened by CT scan of the chest, abdomen, and pelvis for detectable abnormalities or indications of late relapse. Scans are classified as positive or negative, according to standard CT criteria, by a radiologist with expertise in testicular cancer imaging. Patients with negative scans are followed yearly by clinical examination and tumor marker assessment, and every 5 years by CT imaging. Additional follow-up is performed at the discretion of the attending physician. Patients with positive scans undergo confirmation of relapse, whenever possible, by surgical excision or biopsy and treatment is initiated according to best clinical practice. If the follow-up scan is equivocal, patients are advised to have a follow-up scan of the affected region in 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic nonseminomatous germ cell tumor (NSGCT) at risk of developing late relapse of residual abnormality

  * Royal Marsden Hospital stage II-IV disease
* Treatment for NSGCT completed within the past 5 to10 years

  * No evidence of disease after completion of chemotherapy, as demonstrated by negative CT scans within the past 3 years

PATIENT CHARACTERISTICS:

* Willing to attend follow-up for five years
* No contraindication to CT imaging

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-04

PRIMARY OUTCOMES:
Rate of abnormalities due to nonseminomatous germ cell tumour (NSGCT) detected on initial CT-scan

SECONDARY OUTCOMES:
Rate of false positive abnormalities not due to NSGCT but due to benign process
Rate of relapse following initial CT scan
Number of abnormalities detected on second CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Huddart, MD, Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden - Surrey, Sutton, England, United Kingdom